CLINICAL TRIAL: NCT03035838
Title: Importance of Substance P in Intracranial Pressure Elevation Following Traumatic Brain Injury
Acronym: NK1
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Alternate study commenced using different drug
Sponsor: Arun Gupta (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Arun Gupta, Principal Investigator, University of Cambridge
Organization: University of Cambridge (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 212176
Record Dates: First submitted 2017-01-21; First posted 2017-01-30 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — fosaprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Other): There is only one arm in this study. Intracranial pressure and brain swelling will be monitored before and after administration of fosaprepitant
  Interventions: Drug: Fosaprepitant

INTERVENTIONS:
Drug: Fosaprepitant — Within 24 hours from injury, IVAMEND (the intravenous formulation of the NK-1 antagonist fosaprepitant) will be administered at a dose of 300 mg, intravenously over 1 hour.

SUMMARY:
Traumatic brain (TBI) injury is the major cause of morbidity and mortality worldwide especially in population under 40 years of age and has a significant socioeconomic impact. TBI results from the head impacting with an object or from acceleration/deceleration forces that produce vigorous movement of the brain within the skull, with the resultant mechanical forces potentially damaging neurones and blood vessels and causing irreversible, primary brain injury. Primary injury leads to activation of cellular and molecular responses which lead to disruption of the blood-brain barrier causing the brain to swell. As the intracranial space is not expandable (i.e. is fixed), this swelling leads to increase in intracranial pressure (ICP) compromising blood supply to the rest of the brain leading to secondary brain injury. As we are unable to reverse the primary injury, current protocols use supportive measures to control the ICP and ensure optimal blood supply to the brain in an attempt to minimize secondary injury. Our understanding of the factors involved in the initiation and propagation of brain swelling in TBI is growing and the role of neuroinflammatory cytokines in this process is increasingly recognized. In preclinical models of TBI, a specific inflammatory cytokine termed substance P (SP) is found to be associated with blood-brain barrier disruption and development of brain oedema in the immediate phase following injury. The aim of this study is to examine the role of SP in the genesis of cerebral oedema and elevation of ICP and thus secondary injury following human TBI. This would be achieved by blocking SP function with a SP receptor antagonist Fosaprepitant (IVEMEND®, Merck) in the first 24 hours following TBI and then continuously measuring ICP and assessing the evolvement of TBI using magnetic resonance imaging.

DETAILED DESCRIPTION:
All severe traumatic brain injury patients admitted to the Cambridge University Hospital's Neurosciences Critical Care Unit who require insertion of a triple bolt for multimodal neuromonitoring (intracranial pressure-ICP, microdialysis-MD and brain tissue oxygen partial pressure-PbtO2) will be screened for participation in this study. Eligible patients will have an initial MRI scan in the first 24 hours from injury. Following this, and within 24 hours from injury, IVAMEND (the intravenous formulation of the NK-1 antagonist fosaprepitant)will be administered at a dose of 300 mg, intravenously over 1 hour. Patients will then have a follow up MRI scan in the 24 hour following IVAMEND administration. Continuous ICP and PbtO2 monitoring as well as hourly microdialysis sampling will start immediately following insertion of monitors and at least 6 hours before and will continue for at least 12 hours after IVAMEND administration. ICP will continue to be monitored continuously in the 5 days following administration of IVAMEND. Microdialysis samples collected over the period of 6 hours before and 12 hours after the administration of Fosaprepitant will be stored and consequently used to measure the concentration of Substance P, nitric oxide (NO) and inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with traumatic brain injury requiring intracranial pressure monitoring
* Age 18-65 years
* Abnormal CT scan

Exclusion Criteria:

* Bilateral fixed and dilated pupils
* Bleeding diathesis
* Devastating injuries; patient not expected to survive > 24 hours
* Brainstem damage
* Pregnancy
* Sedation with Midazolam
* Patients under 18 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Reduction in intracranial pressure | up to 5 days
  Intracranial pressure will be measured continuously for up to 5 days after intervention

SECONDARY OUTCOMES:
Improvement in brain tissue oxygen tension | up to 5 days
  Brain Tissue Oxygen will be measured continuously for up to 5 days after intervention
Improvement in lactate/pyruvate ratio on microdialysis monitoring | up to 5 days
  Microdialysis will be measured continuously for up to 5 days after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Arun Gupta, MD PhD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No